CLINICAL TRIAL: NCT00814515
Title: A Phase III, Multicenter, Randomized, Controlled, Double-Masked Trial of NOVA22007 (Ciclosporin 0.1%) Ophthalmic Cationic Emulsion Versus Vehicle in Patients With Moderate to Severe Dry Eye Syndrome
Brief Title: Double-Masked Trial of NOVA22007 (Ciclosporin 0.1%) Versus Vehicle in Patients With Moderate to Severe Dry Eye Syndrome
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Santen SAS (Industry)
Responsible Party: Mourad AMRANE, MD, Novagali Pharma
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NVG06C103
Record Dates: First submitted 2008-12-24; First posted 2008-12-25 (Estimated); Last update posted 2010-07-16 (Estimated); Status verified 2010-07

CONDITIONS: Moderate to Severe Dry Eye Syndrome
Keywords: Moderate; Severe; Dry; Eye; Ciclosporin; Cyclosporine
MeSH Terms: conditions — Lymphoma, Follicular

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Ciclosporin 0.1%
  Interventions: Drug: NOVA22007 (Ciclosporin 0.1%)
- 2 (Placebo Comparator): Vehicle
  Interventions: Drug: NOVA22007

INTERVENTIONS:
Drug: NOVA22007 (Ciclosporin 0.1%) — Ciclosporin 0.1% Ophthalmic Emulsions
  Arms: 1
Drug: NOVA22007 — Vehicle
  Arms: 2

SUMMARY:
A Phase III, Multicenter, Randomized, Controlled, Double-Masked Trial of NOVA22007 (Ciclosporin 0.1%) Ophthalmic Cationic Emulsion versus Vehicle in Patients with Moderate to Severe Dry Eye Syndrome

ELIGIBILITY:
Inclusion Criteria:

* Males or females 18 years of age or greater.
* At baseline, moderate to severe dry eye condition persisting despite conventional management.

Exclusion Criteria:

* Presence or history of any systemic or ocular disorder or condition, including ocular surgery, trauma or disease that could possibly interfere with the interpretation of study results.
* Any relevant ocular anomaly interfering with the ocular surface, including post radiation keratitis, Stevens-Johnson syndrome, corneal ulcer history or concomitant corneal ulcer of infectious origin, etc.
* Any other ocular diseases requiring topical ocular treatment during the study period.
* Patient who has participated in a clinical trial with a new active substance during the past month before study entry.
* Participation in another clinical study at the same time as the present study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 482 (Estimated)
Dates: Start 2007-09; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Corneal fluorescein staining (on modified Oxford scale) | Approximately 26 weeks
Patient's global score of all symptoms of ocular discomfort unrelated to study medication instillation, using a visual analog scale (VAS) ranging from 0%-100% | Approximately 26 weeks

SECONDARY OUTCOMES:
• Ocular Symptom Disease Index© (OSDI©) questionnaire • Percentage of complete responder to corneal fluorescein staining (on modified Oxford scale), i.e. with corneal staining score =0 • Patient's score of each symptom of ocular discomfort unrelated to | Approximately 26 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital des XV-XX, Paris, Île-de-France Region, France